CLINICAL TRIAL: NCT00233415
Title: Phase II Study to Evaluate the Efficacy of Conventional Chemoradiotherapy Followed by Stereotactic Radiosurgery for Locally Advanced Pancreatic Cancer
Brief Title: Cyberknife Radiosurgery for Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Albert Koong, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANC0001; NCT00233415; PANC0001
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

INTERVENTIONS:
Device: Stereotactic Radiosurgery (Cyberknife)

SUMMARY:
The purpose of the trial is to test the efficacy of combining conventional chemoradiotherapy with radiosurgery for locally advanced pancreas cancer.

DETAILED DESCRIPTION:
The purpose of the trial is to test the efficacy of treating locally advanced pancreatic cancer with 5FU and concurrent conventional radiotherapy followed by precisely administered single fraction of high-energy radiation using a radiosurgical technique.

ELIGIBILITY:
Inclusion Criteria:- Pancreatic tumors not to exceed 7.5 cm.

* Histologically confirmed malignancies of the pancreas, (ampulla of Vater or periampullary duodenum, tumors may be included when the head of pancreas is secondarily involved and unresectable criteria are met).
* Unresectable by CT criteria or unresectable at exploratory laparotomy or laparoscopy. CT criteria for unresectability include encasement of the superior mesenteric vein (SMV), portal vein (PV) or invasion of the celiac artery or superior mesenteric artery (SMA).
* Patients with metastatic disease may be treated if they are symptomatic from the primary tumor.
* Eastern Clinical Oncology Group performance status 0, 1 or 2. Exclusion Criteria:Chemotherapy within 1 month of registration.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-07; Primary Completion 2006-03 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of Conventional Chemoradiotherapy Followed by Stereotactic Radiosurgery

CONTACTS AND LOCATIONS:
Overall Officials: Albert Koong, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States